CLINICAL TRIAL: NCT02788045
Title: A Randomized, Parallel-Group, Placebo-Controlled, Double-Blind Phase 1/2a Study in Healthy HIV Uninfected Adults to Assess the Safety/Tolerability and Immunogenicity of 2 Different Prime/Boost Regimens; Priming With Trivalent Ad26.Mos.HIV and Boosting With Trivalent Ad26.Mos.HIV And Clade C Gp140 Plus Adjuvant or Priming With Tetravalent Ad26.Mos4.HIV and Boosting With Tetravalent Ad26.Mos4.HIV and Clade C Gp140 Plus Adjuvant
Brief Title: Safety, Tolerability and Immunogenicity Study of Different Vaccine Regimens of Trivalent Ad26.Mos.HIV or Tetravalent Ad26.Mos4.HIV Along With Clade C Glycoprotein (gp)140 in Healthy Human Immunodeficiency Virus (HIV)-Uninfected Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108152; VAC89220HPX2004 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Group 1A: Ad26.Mos.HIV (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12, followed by Ad26.Mos.HIV vaccine + Clade C glycoprotein 140 vaccine containing 250 micrograms (mcg) of total protein mixed with adjuvant (aluminum phosphate) at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: Clade C gp140
- Group 1B: Placebo (Placebo Comparator): Participants will receive placebo at Weeks 0, 12, 24 and 48.
  Interventions: Drug: Placebo
- Group 2A: Ad26.Mos4.HIV (Experimental): Participants will receive Ad26.Mos4.HIV vaccine at Week 0 and 12; followed by Ad26.Mos4.HIV vaccine + Clade C glycoprotein 140 vaccine containing 250 micrograms (mcg) of total protein mixed with adjuvant (aluminum phosphate) at Week 24 and 48. Participants will be included in an optional Long-term Extension (LTE) phase (3 years or 4 years Follow-up after Week 72, every 6 months visit) to assess immunogenicity and safety (serious adverse events [SAEs]).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: Clade C gp140
- Group 2B: Placebo (Placebo Comparator): Participants will receive placebo at Weeks 0, 12, 24 and 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.Mos.HIV — Recombinant replication-deficient Ad26 vectored vaccine and consists of 3 Ad26 vectors, one containing a mosaic insert of envelope (Env) sequence, and 2 vectors containing mosaic inserts of Gag and Pol sequences (Ad26.Mos.1.Env + Ad26.Mos1.Gag-Pol + Ad26.Mos2.Gag-Pol). Total dose is 5*10^10 viral particle per 0.5 milliliter (mL) injection administered intramuscularly.
  Arms: Group 1A: Ad26.Mos.HIV
Biological: Ad26.Mos4.HIV — Recombinant replication-deficient Ad26 vectored vaccine and consists of 4 Ad26 vectors, 2 containing a mosaic insert of envelope (Env) sequence, and 2 vectors containing mosaic inserts of Gag and Pol sequences (Ad26.Mos.1.Env + Ad26.Mos.2S.Env + Ad26.Mos1.Gag-Pol + Ad26.Mos2.Gag-Pol). Total dose is 5*10^10 viral particle per 0.5mL injection administered intramuscularly.
  Arms: Group 2A: Ad26.Mos4.HIV
Biological: Clade C gp140 — Clade C gp140 vaccine containing 250 mcg of total protein, mixed with aluminum phosphate adjuvant, per 0.5 mL injection administered intramuscularly.
  Arms: Group 1A: Ad26.Mos.HIV; Group 2A: Ad26.Mos4.HIV
Drug: Placebo — Normal saline 0.9 percent (%), 0.5 mL injection administered intramuscularly.
  Arms: Group 1B: Placebo; Group 2B: Placebo

SUMMARY:
The purpose of this study is to assess the safety/tolerability of the 2 different vaccine regimens of priming with trivalent Ad26.Mos.HIV and boosting with trivalent Ad26.Mos.HIV and Clade C gp140 plus adjuvant or priming with tetravalent Ad26.Mos4.HIV and boosting with Ad26.Mos4.HIV and Clade C glycoprotein (gp)140 plus adjuvant. Immune responses of the different vaccine schedules will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Are negative for human immunodeficiency virus (HIV) infection at screening
* Is healthy on the basis of physical examination, medical history, electrocardiogram (ECG), and vital signs measurement performed at screening
* Are willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Female participants of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [beta hCG]) at the Screening visit, and a negative urine pregnancy test pre-dose on Day 1
* Are assessed by the clinic staff as being at low risk for HIV infection

Exclusion Criteria:

* Has chronic hepatitis B (measured by hepatitis B surface antigen test) or active hepatitis C (measured by hepatitis C virus [HCV] Ab test; if positive, HCV ribonucleic acid [RNA] PCR test will be used to confirm active versus past HCV infection), active syphilis infection, chlamydia, gonorrhea, or trichomonas . Active syphilis documented by serology unless positive serology is due to past treated infection
* Has had a thyroidectomy or active thyroid disease requiring medication during the last 12 months (not excluded: a stable thyroid supplementation)
* Has had major psychiatric illness and/or substance abuse problems during the past 12 months (including hospitalization or periods of work disability) that in the opinion of the investigator would preclude participation
* Has been in receipt of any licensed vaccine within 14 days prior to the first dose of study vaccine/placebo, plans to receive within 14 days after the first study vaccination, or plans to receive within 14 days before or after the second, third or fourth vaccination
* Is a recipient of a prophylactic or therapeutic HIV vaccine candidate at any time, or a recipient of other experimental vaccine(s) within the last 12 months prior to the Day 1 visit (Vaccination 1). For participants who received an experimental vaccine (except HIV vaccine) more than 12 months prior to the Day 1 visit (Vaccination 1), documentation of the identity of the experimental vaccine must be provided to the sponsor, who will determine eligibility on a case-by-case basis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (10):
- United States (9):
  - Birmingham, Alabama
  - San Francisco, California
  - Decatur, Georgia
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Rochester, New York
  - Philadelphia, Pennsylvania
  - Seattle, Washington
- Kigali, Rwanda

REFERENCES:
- [Derived] Baden LR, Stieh DJ, Sarnecki M, Walsh SR, Tomaras GD, Kublin JG, McElrath MJ, Alter G, Ferrari G, Montefiori D, Mann P, Nijs S, Callewaert K, Goepfert P, Edupuganti S, Karita E, Langedijk JP, Wegmann F, Corey L, Pau MG, Barouch DH, Schuitemaker H, Tomaka F; Traverse/HVTN 117/HPX2004 Study Team. Safety and immunogenicity of two heterologous HIV vaccine regimens in healthy, HIV-uninfected adults (TRAVERSE): a randomised, parallel-group, placebo-controlled, double-blind, phase 1/2a study. Lancet HIV. 2020 Oct;7(10):e688-e698. doi: 10.1016/S2352-3018(20)30229-0. PMID 33010242

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 201 participants were enrolled, out of which 198 participants were randomized and vaccinated; 3 participants were not vaccinated and hence were not included in analyses.
Groups:
- Tetravalent Ad26.Mos4.HIV Vaccine: Participants received adenovirus serotype 26-Mosaic-Human Immunodeficiency Virus (Ad26.Mos4.HIV) vaccine 5*10^10 virus particles (vp) via Intramuscular (IM) injection at Weeks (Wks) 0 and 12. At Weeks 24 and 48, participants received 5*10^10 vp Ad26.Mos4.HIV vaccine and HIV Clade C glycoprotein 140 (gp140) vaccine containing 250 micrograms (mcg) of total protein mixed with adjuvant (aluminum phosphate) as an IM injection. Participants were followed up till Week 72. Participants who had received all 4 vaccinations and were negative for HIV infection at Week 72 were included in an optional Long-term Extension (LTE) phase (up to Week 264).
- Trivalent Ad26.Mos.HIV Vaccine: Participants received Ad26.Mos4.HIV vaccine 5*10^10 vp via IM injection at Weeks 0 and 12. At Weeks 24 and 48 participants received 5*10^10 vp Ad26.Mos.HIV vaccine and HIV Clade C glycoprotein 140 (gp140) vaccine containing 250 mcg of total protein mixed with adjuvant (aluminum phosphate) as an IM injection. Participants were followed up till Week 72.
- Placebo: Participants received placebo matching to either Ad26.Mos4.HIV or Ad26.Mos.HIV as 0.5 mL via IM injection at Weeks 0 and 12, and placebo matching to Clade C gp 140/aluminum phosphate adjuvant as 0.5 mL via IM injection at Weeks 24 and 48. The placebo arms were pooled as there were no differences in the individuals randomized to either of the placebo groups. Participants were followed up till Week 72.
Period: Main Study (Up to Week 72)
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Started | 110 | 55 | 33
Completed | 94 | 45 | 28
Not Completed | 16 | 10 | 5
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 5 | 4 | 3
Not completed — Pregnancy | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 1
Not completed — Other | 3 | 0 | 0
Period: Long Term Extension (From Wk 72 to 264)
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Started | 77 (Only eligible participants entered LTE phase.) | 0 | 0
Completed | 60 | 0 | 0
Not Completed | 17 | 0 | 0
Not completed — Lost to Follow-up | 8 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo | Total
Number analyzed (Participants) | 110 | 55 | 33 | 198
Age, Continuous [Median (Full Range); unit: years] | 28.0 [18 to 50] | 27.0 [19 to 50] | 27.0 [18 to 44] | 27.0 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 32 | 24 | 110
  Male | 56 | 23 | 9 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 4 | 23
  Not Hispanic or Latino | 96 | 48 | 29 | 173
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 5 | 5 | 0 | 10
  Black or African American | 35 | 18 | 7 | 60
  White | 58 | 24 | 23 | 105
  More than one race | 6 | 5 | 2 | 13
  Unknown or Not Reported | 1 | 0 | 1 | 2
  Other | 4 | 2 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  RWANDA | 10 | 5 | 2 | 17
  UNITED STATES | 100 | 50 | 31 | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) Post First Vaccination
Description: Solicited local AEs were predefined local events (at the injection site: erythema, induration, swelling, itching and warmth) that were by definition considered as related to the study vaccine and collected within 7 days after vaccination.
Time Frame: 7 days after first vaccination on Day 1 (Day 8)
Population: The full analysis set (FAS) included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 110 | 55 | 33
percentage of participants | 70.9 | 78.2 | 27.3

2. Primary Outcome: Percentage of Participants With Solicited Local AEs Post Second Vaccination
Description: as for outcome 1
Time Frame: 7 days after second vaccination on Day 85 (Day 92)
Population: The FAS included all participants who were randomized and who received at least one dose of study vaccine. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 102 | 51 | 32
percentage of participants | 83.3 | 76.5 | 50

3. Primary Outcome: Percentage of Participants With Solicited Local AEs Post Third Vaccination
Description: as for outcome 1
Time Frame: 7 days after third vaccination on Day 169 (Day 176)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 99 | 49 | 32
percentage of participants | 80.8 | 79.6 | 21.9

4. Primary Outcome: Percentage of Participants With Solicited Local AEs Post Fourth Vaccination
Description: as for outcome 1
Time Frame: 7 days after fourth vaccination on Day 337 (Day 344)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 94 | 45 | 27
percentage of participants | 84 | 68.9 | 29.6

5. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Post First Vaccination
Description: An AE was defined as any untoward medical event that occurred in a participant administered an investigational product, and it did not necessarily indicated only events with clear causal relationship with the relevant investigational product. Solicited systemic AEs including pyrexia/fever, headache, fatigue, myalgia, nausea and chills were collected within 7 days after vaccination.
Time Frame: 7 days after first vaccination on Day 1 (Day 8)
Population: FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 110 | 55 | 33
percentage of participants | 69.1 | 83.6 | 54.5

6. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Post Second Vaccination
Description: as for outcome 5
Time Frame: 7 days after second vaccination on Day 85 (Day 92)
Population: FAS included all participants who were randomized and who received at least one dose of study vaccine. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 102 | 51 | 32
percentage of participants | 66.7 | 54.9 | 40.6

7. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Post Third Vaccination
Description: as for outcome 5
Time Frame: 7 days after third vaccination on Day 169 (Day 176)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 99 | 49 | 32
percentage of participants | 59.6 | 44.9 | 34.4

8. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Post Fourth Vaccination
Description: as for outcome 5
Time Frame: 7 days after fourth vaccination on Day 337 (Day 344)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 94 | 45 | 27
percentage of participants | 58.5 | 53.3 | 33.3

9. Primary Outcome: Percentage of Participants With Unsolicited AEs for 28 Days After First Vaccination
Description: An AE was defined as any untoward medical event that occurred in a participant administered an investigational product, and it did not necessarily indicated only events with clear causal relationship with the relevant investigational product. Unsolicited AEs were defined as the AEs other than those categorized as "solicited AEs" and were required to be collected for any events that occurred from the time of vaccination and through the subsequent 28 days.
Time Frame: 28 days after first vaccination on Day 1 (Day 29)
Population: The FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 110 | 55 | 33
percentage of participants | 38.2 | 41.8 | 30.3

10. Primary Outcome: Percentage of Participants With Unsolicited AEs for 28 Days After Second Vaccination
Description: as for outcome 9
Time Frame: 28 days after second vaccination on Day 85 (Day 113)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 102 | 51 | 32
percentage of participants | 30.4 | 23.5 | 37.5

11. Primary Outcome: Percentage of Participants With Unsolicited AEs for 28 Days After Third Vaccination
Description: as for outcome 9
Time Frame: 28 days after third vaccination on Day 169 (Day 197)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 99 | 49 | 32
percentage of participants | 28.3 | 20.4 | 21.9

12. Primary Outcome: Percentage of Participants With Unsolicited AEs for 28 Days After Fourth Vaccination
Description: as for outcome 9
Time Frame: 28 days after fourth vaccination on Day 334 (Day 362)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 94 | 45 | 27
percentage of participants | 36.2 | 22.2 | 40.7

13. Primary Outcome: Percentage of Participants With Discontinuations From Vaccination Due to AEs
Description: Percentage of participants with discontinuations from vaccination due to AEs were reported.
Time Frame: Up to Week 72
Population: The FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 110 | 55 | 33
percentage of participants | 0 | 1.8 | 6.1

14. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) During Main Study
Description: An AE was defined as any untoward medical event that occurred in a participant administered an investigational product, and it did not necessarily indicated only events with clear causal relationship with the relevant investigational product. SAE was defined as any AE that resulted in: death, persistent or significant disability/incapacity, required inpatient hospitalization or prolongation of existing hospitalization, was life-threatening experience, was a congenital anomaly/birth defect and would jeopardize participant and/or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Week 72
Population: The FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 110 | 55 | 33
percentage of participants | 5.5 | 0 | 0

15. Primary Outcome: Percentage of Participants With SAEs During Long Term Extension (LTE) Period
Description: An AE was defined as any untoward medical event that occurred in a participant administered an investigational product, and it did not necessarily indicated only events with clear causal relationship with the relevant investigational product. SAE was defined as any AE that resulted in: death, persistent or significant disability/incapacity, required inpatient hospitalization or prolongation of existing hospitalization, was life-threatening experience, was a congenital anomaly/birth defect and would jeopardize participant and/or required medical or surgical intervention to prevent one of the outcomes listed above. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: From Week 96 to Week 264
Population: The FAS included all participants those were all the participants from the Tetravalent Ad26.Mos4.HIV group who had received all 4 vaccinations and were negative for HIV infections at Week 72.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine
Number analyzed (Participants) | 77
percentage of participants | 5.2

16. Primary Outcome: Percentage of Participants With AEs of Special Interest During Main Study
Description: Percentage of participants with AEs of special interest during main study were reported. HIV infection was considered as an AE of special interest.
Time Frame: Up to Week 72
Population: The FAS included all participants who were randomized and who received at least one dose of study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 110 | 55 | 33
percentage of participants | 0 | 0 | 0

17. Primary Outcome: Percentage of Participants With AEs of Special Interest During LTE Period
Description: Percentage of participants with AEs of special interest during LTE period were reported. HIV infection was considered as an AE of special interest. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: From Week 96 to Week 264
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine
Number analyzed (Participants) | 77
percentage of participants | 0

18. Primary Outcome: Percentage of Responders for Envelop (Env) Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012) Specific Binding Antibody Titers at Week 28
Description: Percentage of responders for envelop (Env) Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012) specific binding antibody titers at Week 28 were reported. Env Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012)-specific binding antibody titers were assessed using enzyme-linked immunosorbent assay (ELISA). The response was defined as post-baseline value greater than (>) lower limit of quantification (LLOQ) if baseline value less than (<) LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline value greater than or equal to (>=) LLOQ.
Time Frame: Week 28
Population: The PPI analysis set included all participants who had received at least first three vaccinations, according to protocol-specified vaccination schedule (+/- 2 weeks), had at least 1 measured post-dose blood sample collected and were not diagnosed with HIV infection during the study. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure; 'n' (number analyzed) signifies number of participants evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 98 | 48 | 31
percentage of responders
  Clade A (92UG037.1) | 100 [96.3 to 100.0] | 100 [92.6 to 100.0] | 19.4 [7.5 to 37.5]
  Clade B (1990a) | 100 [96.3 to 100.0] | 100 [92.6 to 100.0] | 12.9 [3.6 to 29.8]
  Clade C (Con C): number analyzed (Participants) | 96 | 48 | 31
  Clade C (Con C) | 100 [96.2 to 100] | 100 [92.6 to 100] | 12.9 [3.6 to 29.8]
  Clade C (C97ZA.012) | 100 [96.3 to 100] | 100 [92.6 to 100] | 6.5 [0.8 to 21.4]

19. Primary Outcome: Percentage of Responders for Envelop (Env) Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012) Specific Binding Antibody Titers at Week 52
Description: Percentage of responders for envelop (Env) Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012) specific binding antibody titers at Week 52 were reported. Env Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012)-specific binding antibody titers were assessed using enzyme-linked immunosorbent assay (ELISA). The response was defined as post-baseline value greater than (>) lower limit of quantification (LLOQ) if baseline value less than (<) LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline value greater than or equal to (>=) LLOQ.
Time Frame: Week 52
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 98 | 48 | 31
percentage of responders
  Clade A (92UG037.1): number analyzed (Participants) | 93 | 40 | 27
  Clade A (92UG037.1) | 100 [96.1 to 100.0] | 100 [91.2 to 100.0] | 0 [0 to 0]
  Clade B (1990a): number analyzed (Participants) | 93 | 40 | 27
  Clade B (1990a) | 100 [96.1 to 100] | 100 [91.2 to 100] | 22.2 [8.6 to 42.3]
  Clade C (Con C): number analyzed (Participants) | 93 | 40 | 27
  Clade C (Con C) | 100 [96.1 to 100] | 100 [91.2 to 100] | 0 [0 to 0]
  Clade C (C97ZA.012): number analyzed (Participants) | 93 | 40 | 27
  Clade C (C97ZA.012) | 100 [96.1 to 100] | 100 [91.2 to 100] | 3.7 [0.1 to 19.0]

20. Primary Outcome: Percentage of Responders for Envelop (Env) Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012) Specific Binding Antibody Titers at Week 72
Description: Percentage of responders for envelop (Env) Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012) specific binding antibody titers at Week 72 were reported. Env Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012)-specific binding antibody titers were assessed using enzyme-linked immunosorbent assay (ELISA). The response was defined as post-baseline value greater than (>) lower limit of quantification (LLOQ) if baseline value less than (<) LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline value greater than or equal to (>=) LLOQ.
Time Frame: Week 72
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 98 | 48 | 31
percentage of responders
  Clade A (92UG037.1): number analyzed (Participants) | 92 | 43 | 27
  Clade A (92UG037.1) | 100 [96.1 to 100.0] | 100 [91.8 to 100.0] | 2 [0.9 to 24.3]
  Clade B (1990a): number analyzed (Participants) | 92 | 43 | 27
  Clade B (1990a) | 100 [96.1 to 100] | 100 [91.8 to 100] | 11.1 [2.4 to 29.2]
  Clade C (Con C): number analyzed (Participants) | 91 | 43 | 27
  Clade C (Con C) | 100 [96 to 100] | 100 [91.8 to 100] | 0 [0 to 0]
  Clade C (C97ZA.012): number analyzed (Participants) | 92 | 43 | 27
  Clade C (C97ZA.012) | 100 [96.1 to 100] | 100 [91.8 to 100] | 3.7 [0.1 to 19]

21. Secondary Outcome: Percentage of Responders for Human Immunodeficiency Virus Neutralizing Antibody (HIV nAb)
Description: The functionality of vaccine-induced antibody responses was investigated by the determination of nAb activity in a virus neutralization assay (VNA) using TZM-bl cells and Env-pseudotyped viruses. The response was defined as post-baseline value >LLOQ. The LLOQ for this assay was an inhibitory concentration (IC50) of 20 (fold-dilution). The data was collected for the responses against Tier 1 HIV strain Clade C (MW965.26 and C97ZA.012).
Time Frame: Weeks 28, 52 and 72
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 98 | 48 | 30
percentage of responders
  Clade C (MW965.26) Week 28 | 99 [94.4 to 100.0] | 66.7 [51.6 to 79.6] | 0 [0 to 0]
  Clade C (MW965.26) Week 52: number analyzed (Participants) | 93 | 40 | 27
  Clade C (MW965.26) Week 52 | 100 [96.1 to 100.0] | 90 [76.3 to 97.2] | 0 [0 to 0]
  Clade C (MW965.26) Week 72: number analyzed (Participants) | 94 | 24 | 0
  Clade C (MW965.26) Week 72 | 98.9 [94.1 to 100.0] | 100 [85.8 to 100.0] |
  Clade C (C97ZA.012) Week 28 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Clade C (C97ZA.012) Week 52: number analyzed (Participants) | 93 | 40 | 27
  Clade C (C97ZA.012) Week 52 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

22. Secondary Outcome: Percentage of Responders for Env Antibody-dependent Cellular Phagocytosis (ADCP) gp Antibody
Description: The functionality of vaccine-induced antibody responses was investigated by the determination of ADCP. The response was defined as post-baseline value > limit of detection (LOD) if baseline value <LOD or missing or defined as post-baseline value >3-fold increase from baseline if baseline value >=LOD. The lower limits of detection (LODs) for this assay were 5.16, 6.43, 6.49, 4.32 and 4.28 (phagocytic score) for Clade A (92UG037.1), Clade B (1990a), Clade C (Con C), Clade C (C97ZA.012), and Mos1, respectively.
Time Frame: Weeks 28, 52 and 72
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 98 | 47 | 31
percentage of responders
  Clade A (92UG037.1) at Week 28 | 72.4 [62.5 to 81] | 36.2 [22.7 to 51.5] | 0 [0 to 0]
  Clade B (1990a) at Week 28 | 69.4 [59.3 to 78.3] | 57.4 [42.2 to 71.7] | 0 [0 to 0]
  Clade C (Con C) at Week 28 | 88.8 [80.8 to 94.3] | 66 [50.7 to 79.1] | 16.1 [5.5 to 33.7]
  Mos1 at Week 28 | 100 [96.3 to 100] | 100 [92.5 to 100] | 0 [0 to 0]
  Clade C (C97ZA.012) at Week 28 | 98 [92.8 to 99.8] | 93.6 [82.5 to 98.7] | 3.2 [0.1 to 16.7]
  Clade C (C97ZA.012) at Week 52: number analyzed (Participants) | 93 | 40 | 27
  Clade C (C97ZA.012) at Week 52 | 97.8 [92.4 to 99.7] | 82.5 [67.2 to 92.7] | 0 [0 to 0]
  Clade C (C97ZA.012) at Week 72: number analyzed (Participants) | 92 | 43 | 27
  Clade C (C97ZA.012) at Week 72 | 98.9 [94.1 to 100] | 97.7 [87.7 to 99.9] | 18.5 [6.3 to 38.1]

23. Secondary Outcome: Percentage of Responders With Interferon-gamma (IFN-gamma) T Cell Responses Assessed Using Enzyme-linked Immunospot Assay (ELISpot)
Description: Frozen peripheral blood mononuclear cell (PBMCs) were analyzed by interferon-gamma (IFN-gamma) (ELISpot). The response was defined as post-baseline value >P95 if baseline <P95 or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=P95.
Time Frame: Weeks 26, 52 and 72
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 99 | 48 | 31
percentage of responders
  ENV peptide pool potential T-cell epitope (PTE) at Week 26 | 96 [90.0 to 98.9] | 79.2 [65 to 89.5] | 3.2 [0.1 to 16.7]
  ENV peptide pool PTE at Week 52: number analyzed (Participants) | 92 | 40 | 26
  ENV peptide pool PTE at Week 52 | 95.7 [89.2 to 98.8] | 85 [70.2 to 94.3] | 3.8 [0.1 to 19.6]
  ENV peptide pool PTE at Week 72: number analyzed (Participants) | 89 | 42 | 27
  ENV peptide pool PTE at Week 72 | 97.8 [92.1 to 99.7] | 83.3 [68.6 to 93] | 3.7 [0.1 to 19]
  ENV peptide pool Mos1 at Week 26 | 96 [90 to 98.9] | 87.5 [74.8 to 95.3] | 6.5 [0.8 to 21.4]
  ENV peptide pool Mos1 at Week 52: number analyzed (Participants) | 92 | 40 | 26
  ENV peptide pool Mos1 at Week 52 | 98.9 [94.1 to 100] | 92.5 [79.6 to 98.4] | 3.8 [0.1 to 19.6]
  ENV peptide pool Mos1 at Week 72: number analyzed (Participants) | 89 | 42 | 27
  ENV peptide pool Mos1 at Week 72 | 97.8 [92.1 to 99.7] | 92.9 [80.5 to 98.5] | 18.5 [6.3 to 38.1]
  ENV peptide pool Mos2 at Week 26 | 96 [90 to 98.9] | 58.3 [43.2 to 72.4] | 3.2 [0.1 to 16.7]
  ENV peptide pool Mos2 at Week 52: number analyzed (Participants) | 92 | 40 | 26
  ENV peptide pool Mos2 at Week 52 | 93.5 [86.3 to 97.6] | 77.5 [61.5 to 89.2] | 3.8 [0.1 to 19.6]
  ENV peptide pool Mos2 at Week 72: number analyzed (Participants) | 89 | 40 | 27
  ENV peptide pool Mos2 at Week 72 | 95.5 [88.9 to 98.8] | 70 [53.5 to 83.4] | 0 [0 to 0]
  Gag peptide pool PTE at Week 26 | 58.6 [48.2 to 68.4] | 60.4 [45.3 to 74.2] | 3.2 [0.1 to 16.7]
  Gag peptide pool PTE at Week 52: number analyzed (Participants) | 92 | 40 | 26
  Gag peptide pool PTE at Week 52 | 57.6 [46.9 to 67.9] | 70 [53.5 to 83.4] | 0 [0 to 0]
  Gag peptide pool PTE at Week 72: number analyzed (Participants) | 89 | 42 | 27
  Gag peptide pool PTE at Week 72 | 41.6 [31.2 to 52.5] | 47.6 [32 to 63.6] | 0 [0 to 0]
  Gag peptide pool Mos1 at Week 26 | 59.6 [49.3 to 69.3] | 54.2 [39.2 to 68.6] | 0 [0 to 0]
  Gag peptide pool Mos1 at Week 52: number analyzed (Participants) | 92 | 40 | 26
  Gag peptide pool Mos1 at Week 52 | 60.9 [50.1 to 70.9] | 60 [43.3 to 75.1] | 3.8 [0.1 to 19.6]
  Gag peptide pool Mos1 at Week 72: number analyzed (Participants) | 89 | 42 | 27
  Gag peptide pool Mos1 at Week 72 | 57.3 [46.4 to 67.7] | 54.8 [38.7 to 70.2] | 3.7 [0.1 to 19]
  Gag peptide pool Mos2 at Week 26 | 69.7 [59.6 to 78.5] | 60.4 [45.3 to 74.2] | 0 [0 to 0]
  Gag peptide pool Mos2 at Week 52: number analyzed (Participants) | 92 | 40 | 26
  Gag peptide pool Mos2 at Week 52 | 65.2 [54.6 to 74.9] | 62.5 [45.8 to 77.3] | 0 [0 to 0]
  Gag peptide pool Mos2 at Week 72: number analyzed (Participants) | 89 | 40 | 27
  Gag peptide pool Mos2 at Week 72 | 64 [53.2 to 73.9] | 60 [43.3 to 75.1] | 0 [0 to 0]
  Pol peptide pool PTE at Week 26 | 87.9 [79.8 to 93.6] | 91.7 [80 to 97.7] | 0 [0 to 0]
  Pol peptide pool PTE at Week 52: number analyzed (Participants) | 92 | 40 | 26
  Pol peptide pool PTE at Week 52 | 84.8 [75.8 to 91.4] | 85 [70.2 to 94.3] | 3.8 [0.1 to 19.6]
  Pol peptide pool PTE at Week 72: number analyzed (Participants) | 89 | 40 | 27
  Pol peptide pool PTE at Week 72 | 87.6 [79 to 93.7] | 90 [76.3 to 97.2] | 11.1 [2.4 to 29.2]
  Pol peptide pool Mos1 at Week 26 | 88.9 [81.0 to 94.3] | 85.4 [72.2 to 93.9] | 3.2 [0.1 to 16.7]
  Pol peptide pool Mos1 at Week 52: number analyzed (Participants) | 92 | 40 | 26
  Pol peptide pool Mos1 at Week 52 | 82.6 [73.3 to 89.7] | 92.5 [79.6 to 98.4] | 3.8 [0.1 to 19.6]
  Pol peptide pool Mos1 at Week 72: number analyzed (Participants) | 89 | 42 | 27
  Pol peptide pool Mos1 at Week 72 | 85.4 [76.3 to 92.0] | 81 [65.9 to 91.4] | 14.8 [4.2 to 33.7]
  Pol peptide pool Mos2 at Week 26 | 92.9 [86 to 97.1] | 93.8 [82.8 to 98.7] | 3.2 [0.1 to 16.7]
  Pol peptide pool Mos2 at Week 52: number analyzed (Participants) | 92 | 40 | 26
  Pol peptide pool Mos2 at Week 52 | 89.1 [80.9 to 94.7] | 90 [76.3 to 97.2] | 3.8 [0.1 to 19.6]
  Pol peptide pool Mos2 at Week 72: number analyzed (Participants) | 89 | 40 | 27
  Pol peptide pool Mos2 at Week 72 | 89.9 [81.7 to 95.3] | 92.5 [79.6 to 98.4] | 7.4 [0.9 to 24.3]

24. Secondary Outcome: Percentage of Responders for Immunoglobulin G1 (IgG1) and IgG3 Gylcoprotein (gp) 140 Binding Antibody Assessed Using Clade C (C97ZA.012) Env Enzyme-linked Immunosorbent Assay (ELISA)
Description: Vaccine-induced binding antibody IgG1 and IgG3 subclass responses were investigated using Clade C (C97ZA.012) specific ELISAs. The response was defined as post-baseline value >LLOQ if baseline <LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LLOQ. The LLOQs for this assay were 12.3 and 12.4 for IgG1 and IgG3, respectively.
Time Frame: Weeks 28, 52 and 72
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 93 | 44 | 29
percentage of responders
  Clade C (C97ZA.012) IgG1 at Week 28: number analyzed (Participants) | 92 | 44 | 29
  Clade C (C97ZA.012) IgG1 at Week 28 | 72.8 [62.6 to 81.6] | 61.4 [45.5 to 75.6] | 0 [0 to 0]
  Clade C (C97ZA.012) IgG1 at Week 52: number analyzed (Participants) | 93 | 40 | 27
  Clade C (C97ZA.012) IgG1 at Week 52 | 73.1 [62.9 to 81.8] | 67.5 [50.9 to 81.4] | 0 [0 to 0]
  Clade C (C97ZA.012) IgG1 at Week 72: number analyzed (Participants) | 91 | 42 | 27
  Clade C (C97ZA.012) IgG1 at Week 72 | 67.0 [56.4 to 76.5] | 50 [34.2 to 65.8] | 0 [0 to 0]
  Clade C (C97ZA.012) IgG3 at Week 28: number analyzed (Participants) | 92 | 44 | 29
  Clade C (C97ZA.012) IgG3 at Week 28 | 67.4 [56.8 to 76.8] | 18.2 [8.2 to 32.7] | 0 [0 to 0]
  Clade C (C97ZA.012) IgG3 at Week 52: number analyzed (Participants) | 92 | 39 | 27
  Clade C (C97ZA.012) IgG3 at Week 52 | 66.3 [55.7 to 75.8] | 46.2 [30.1 to 62.8] | 0 [0 to 0]
  Clade C (C97ZA.012) IgG3 at Week 72: number analyzed (Participants) | 89 | 42 | 22
  Clade C (C97ZA.012) IgG3 at Week 72 | 37.1 [27.1 to 48] | 31 [17.6 to 47.1] | 0 [0 to 0]

25. Secondary Outcome: Percentage of Responders for CD4+ and CD8+ T-Cell Responses
Description: Intracellular cytokine staining (ICS) was performed to examine the type of T-cell responding to vaccination. Responder definition was based on the Fisher's exact text between cytokine producing cells and non-producing cells in stimulated versus non-stimulated conditions.
Time Frame: Weeks 28, 52 and 72
Population: The PPI analysis set included all participants who had received at least first three vaccinations, according to protocol-specified vaccination schedule (+/- 2 weeks), had at least 1 measured post-dose blood sample collected and were not diagnosed with HIV during the study. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure; 'n' (number analyzed) signifies number of participants evaluable at specified categories
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 97 | 48 | 31
percentage of responders
  CD4+ ENV pep pool (PP) (Mos1) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 52 | 20 | 1
  CD4+ ENV pep pool (PP) (Mos1) IFNg+ /IL2+ Wk 28 | 53.61 [43.19 to 63.80] | 41.67 [27.61 to 56.79] | 3.23 [0.08 to 16.70]
  CD4+ ENV PP (Mos1) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 59 | 20 | 0
  CD4+ ENV PP (Mos1) IFNg+ /IL2+ Wk 52 | 64.84 [54.12 to 74.56] | 50.00 [33.80 to 66.20] |
  CD4+ ENV PP (Mos1) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 42 | 14 | 0
  CD4+ ENV PP (Mos1) IFNg+ /IL2+ Wk 72 | 53.85 [42.18 to 65.21] | 36.84 [21.81 to 54.01] |
  CD4+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 55 | 21 | 1
  CD4+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 28 | 56.70 [46.25 to 66.73] | 43.75 [29.48 to 58.82] | 3.23 [0.08 to 16.70]
  CD4+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 69 | 22 | 0
  CD4+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 52 | 75.82 [65.72 to 84.19] | 55 [38.49 to 70.74] |
  CD4+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 50 | 14 | 0
  CD4+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 72 | 64.10 [52.44 to 74.66] | 36.84 [21.81 to 54.01] |
  CD4+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 45 | 9 | 0
  CD4+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 28 | 46.39 [36.20 to 56.81] | 18.75 [8.95 to 32.63] |
  CD4+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 58 | 14 | 0
  CD4+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 52 | 63.74 [52.99 to 73.56] | 35.00 [20.63 to 51.68] |
  CD4+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 40 | 4 | 0
  CD4+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 72 | 51.28 [39.69 to 62.77] | 10.53 [2.94 to 24.80] |
  CD4+ ENV pol gag PP IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 56 | 22 | 1
  CD4+ ENV pol gag PP IFNg+ /IL2+ Wk 28 | 57.73 [47.28 to 67.70] | 45.83 [31.37 to 60.83] | 3.23 [0.08 to 16.70]
  CD4+ ENV pol gag PP IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 69 | 22 | 0
  CD4+ ENV pol gag PP IFNg+ /IL2+ Wk 52 | 75.82 [65.72 to 84.19] | 55 [38.49 to 70.74] |
  CD4+ ENV pol gag PP IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 50 | 14 | 0
  CD4+ ENV pol gag PP IFNg+ /IL2+ Wk 72 | 64.10 [52.44 to 74.66] | 36.84 [21.81 to 54.01] |
  CD4+ ENV gag PP ANY IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 8 | 3 | 0
  CD4+ ENV gag PP ANY IFNg+ /IL2+ Wk 28 | 8.25 [3.63 to 15.61] | 6.25 [1.31 to 17.20] |
  CD4+ ENV gag PP ANY IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 3 | 4 | 0
  CD4+ ENV gag PP ANY IFNg+ /IL2+ Wk 52 | 3.30 [0.69 to 9.33] | 10.00 [2.79 to 23.66] |
  CD4+ ENV gag PP ANY IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 2 | 2 | 0
  CD4+ ENV gag PP ANY IFNg+ /IL2+ Wk 72 | 2.56 [0.31 to 8.96] | 5.26 [0.64 to 17.75] |
  CD4+ ENV Pol PP (Mos1) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 8 | 4 | 0
  CD4+ ENV Pol PP (Mos1) IFNg+ /IL2+ Wk 28 | 8.25 [3.63 to 15.61] | 8.33 [2.32 to 19.98] |
  CD4+ ENV Pol PP (Mos1) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 6 | 3 | 0
  CD4+ ENV Pol PP (Mos1) IFNg+ /IL2+ Wk 52 | 6.59 [2.46 to 13.80] | 7.50 [1.57 to 20.39] |
  CD4+ ENV Pol PP (Mos1) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 5 | 2 | 0
  CD4+ ENV Pol PP (Mos1) IFNg+ /IL2+ Wk 72 | 6.41 [2.11 to 14.33] | 5.26 [0.64 to 17.75] |
  CD8+ ENV PP (Mos1) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 34 | 21 | 0
  CD8+ ENV PP (Mos1) IFNg+ /IL2+ Wk 28 | 35.42 [25.92 to 45.84] | 43.75 [29.48 to 58.82] |
  CD8+ ENV PP (Mos1) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 28 | 17 | 0
  CD8+ ENV PP (Mos1) IFNg+ /IL2+ Wk 52 | 30.77 [21.51 to 41.32] | 42.50 [27.04 to 59.11] |
  CD8+ ENV PP (Mos1) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 23 | 10 | 0
  CD8+ ENV PP (Mos1) IFNg+ /IL2+ Wk 72 | 29.11 [19.43 to 40.42] | 26.32 [13.40 to 43.10] |
  CD8+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 40 | 22 | 0
  CD8+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 28 | 41.67 [31.68 to 52.18] | 45.83 [31.37 to 60.83] |
  CD8+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 31 | 18 | 0
  CD8+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 52 | 34.07 [24.45 to 44.75] | 45.00 [29.26 to 61.51] |
  CD8+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 27 | 11 | 0
  CD8+ ENV PP (Mos1 ZA PTE) IFNg+ /IL2+ Wk 72 | 34.18 [23.87 to 45.71] | 28.95 [15.42 to 45.90] |
  CD8+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 21 | 11 | 31
  CD8+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 28 | 21.88 [14.08 to 31.47] | 22.92 [12.03 to 37.31] | 0 [0 to 0]
  CD8+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 14 | 7 | 0
  CD8+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 52 | 15.38 [8.67 to 24.46] | 17.50 [7.34 to 32.78] |
  CD8+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 13 | 4 | 0
  CD8+ ENV PP clade C (ZA) IFNg+ /IL2+ Wk 72 | 16.46 [9.06 to 26.49] | 10.53 [2.94 to 24.80] |
  CD8+ ENV Pol gag PP IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 73 | 39 | 1
  CD8+ ENV Pol gag PP IFNg+ /IL2+ Wk 28 | 76.04 [66.25 to 84.17] | 81.25 [67.37 to 91.05] | 3.23 [0.08 to 16.70]
  CD8+ ENV Pol gag PP IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 65 | 31 | 1
  CD8+ ENV Pol gag PP IFNg+ /IL2+ Wk 52 | 71.43 [61.00 to 80.41] | 77.50 [61.55 to 89.16] | 3.70 [0.09 to 18.97]
  CD8+ ENV Pol gag PP IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 55 | 25 | 1
  CD8+ ENV Pol gag PP IFNg+ /IL2+ Wk 72 | 69.62 [58.25 to 79.47] | 65.79 [48.65 to 80.37] | 4.00 [0.10 to 20.35]
  CD8+ ENV gag PP ANY IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 38 | 19 | 1
  CD8+ ENV gag PP ANY IFNg+ /IL2+ Wk 28 | 39.58 [29.75 to 50.08] | 39.58 [25.77 to 54.73] | 3.23 [0.08 to 16.70]
  CD8+ ENV gag PP ANY IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 29 | 13 | 1
  CD8+ ENV gag PP ANY IFNg+ /IL2+ Wk 52 | 32.91 [22.75 to 44.40] | 31.58 [17.50 to 48.65] | 4.00 [0.10 to 20.35]
  CD8+ Pol PP (Mos1) IFNg+ /IL2+ Wk 28: number analyzed (Participants) | 60 | 30 | 0
  CD8+ Pol PP (Mos1) IFNg+ /IL2+ Wk 28 | 62.50 [52.03 to 72.18] | 62.50 [47.35 to 76.05] |
  CD8+ Pol PP (Mos1) IFNg+ /IL2+ Wk 52: number analyzed (Participants) | 50 | 20 | 0
  CD8+ Pol PP (Mos1) IFNg+ /IL2+ Wk 52 | 54.95 [44.16 to 65.40] | 50.00 [33.80 to 66.20] |
  CD8+ Pol PP (Mos1) IFNg+ /IL2+ Wk 72: number analyzed (Participants) | 41 | 14 | 0
  CD8+ Pol PP (Mos1) IFNg+ /IL2+ Wk 72 | 51.90 [40.36 to 63.29] | 36.84 [21.81 to 54.01] |

26. Secondary Outcome: Percentage of Participants With T-cell Development
Description: As per change in planned analysis, this outcome measure was not performed since it was no longer considered relevant to interpret the immunogenicity of the vaccines.
Time Frame: Up to Week 264
Population: The PPI analysis set included all participants who had received at least first three vaccinations, according to protocol-specified vaccination schedule (+/- 2 weeks), had at least 1 measured post-dose blood sample collected and were not diagnosed with HIV infection during the study.
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 264
Description: The full analysis set (FAS) included of all participants who were randomized and who received atleast one dose of study vaccine. One participant had serious adverse event during main study and long-term extension period. This participant has only been counted once in the adverse event section
Arm/Group | Tetravalent Ad26.Mos4.HIV Vaccine | Trivalent Ad26.Mos.HIV Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/55 | 0/33
Serious Adverse Events (participants affected / at risk) | 9/110 | 0/55 | 0/33
Other Adverse Events (participants affected / at risk) | 37/110 | 22/55 | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tetravalent Ad26.Mos4.HIV Vaccine (N=110) | Trivalent Ad26.Mos.HIV Vaccine (N=55) | Placebo (N=33)
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acoustic Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Bipolar I Disorder (Psychiatric disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tetravalent Ad26.Mos4.HIV Vaccine (N=110) | Trivalent Ad26.Mos.HIV Vaccine (N=55) | Placebo (N=33)
Gastroenteritis (Infections and infestations) | 5 | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 9 | 10
Urinary Tract Infection (Infections and infestations) | 2 | 4 | 0
Viral Infection (Infections and infestations) | 7 | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 5 | 2 | 3
Haemoglobin Decreased (Investigations) | 0 | 3 | 0
Proteinuria (Renal and urinary disorders) | 3 | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2

LIMITATIONS AND CAVEATS:
In this study, the ability to generalize the study outcomes is limited to populations that were included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT02788045/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT02788045/SAP_001.pdf